CLINICAL TRIAL: NCT05705154
Title: Connecting Breath and Mind: Development of an Online Holistic Treatment Programme Connecting Psychological Wellbeing and Breathing Techniques in Children and Young People With Long COVID
Brief Title: Connecting Breath and Mind for CYP With Long COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 315063
Record Dates: First submitted 2022-12-15; First posted 2023-01-30 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Post-COVID-19 Syndrome; Anxiety; Breathlessness
Keywords: Teenager; Adolescent
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Anxiety Disorders; Dyspnea

STUDY DESIGN:
Intervention Model Description: Participants will be randomised using block randomisation into either standard intervention arm or standard intervention plus the new co-designed intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Standard treatment consists of virtual MDT discussion with referrer and advice signposting into local services for specific issues. If a patient is severely affected enough to be seen face to face, they are offered an interdisciplinary consultation, and tailored input from PT OT and psychological services.
  Access to standardised information covering the following topics: sleep, pacing, activity management, school reintegration, managing friendships, eating well and emotional wellbeing.
  More complex or severely affected patients will receive one to one treatment with members of the MDT as required.
  Interventions: Behavioral: Psychology interventions
- Intervention (Experimental): As above standard intervention plus the new co-designed intervention.
  Based on clinical expertise and theory, it is anticipated the following elements may be included in the intervention:
  * Progressive breathing pattern retraining, including education, self-observation, relaxation, body scanning, postural re-alignment
  * Identifying the connections between body and mind to address anxiety and breathlessness
  * Coping skills for managing anxiety using principles from narrative therapy and mindfulness
  * Online materials to improve self-efficacy with home practice
  * Social connection with other CYP for peer support, and resource sharing
  * Activities to help CYP reconnect with their usual activities, skills, abilities, interests, support systems.
  Interventions: Behavioral: Psychology interventions

INTERVENTIONS:
Behavioral: Psychology interventions — Based on clinical expertise and theory, it is anticipated the following elements may be included in the intervention:
  * Progressive breathing pattern retraining, including education, self-observation, relaxation, body scanning, postural re-alignment
  * Identifying the connections between body and mind to address anxiety and breathlessness
  * Coping skills for managing anxiety using principles from narrative therapy and mindfulness
  * Online materials to improve self-efficacy with home practice
  * Social connection with other CYP for peer support, and resource sharing
  * Activities to help CYP reconnect with their usual activities, skills, abilities, interests, support systems.
  Other Names: breathing pattern retraining

SUMMARY:
Recruitment target: Phase I: Co-design of intervention: 5 to 15 CYP aged between 12-18 years of age referred to the pan-London long COVID MDT.

Phase II: Randomised pilot: 40 patients (12-18 years) will be recruited from a potential pool of 214 patients referred to the pan-London long COVID MDT.

Methods: Phase I: Co-design Design and setting The intervention will be co-designed with CYP following a process informed by practice-base evidence, which centres the voices and wisdom of CYP, focuses on creativity and playfulness, and systemic and narrative approaches. The process will involve: 1) Refining the intentions of key stakeholders (including ways of bringing psychological and physiological principles into the intervention); 2) Participation of CYP; 3) Creativity and playfulness and 4) Responding to feedback (see Salvo et al., 2022).

Phase II. Pilot Population: 40 patients (12-18 years) will be recruited from a potential pool of 214 patients referred to the pan-London long COVID MDT. CYP will be randomised to receive either standard treatment or standard treatment plus intervention.

Study Treatment Standard treatment consists of virtual MDT discussion with referrer and advice signposting into local services for specific issues. They are sent leaflets and information. If a patient is severely affected enough to be seen face to face, they are offered an interdisciplinary consultation, and tailored input from therapies and psychological services.

Access to bite size videos and leaflets covering the following topics: sleep, pacing, activity management, school reintegration, managing friendships, eating well and emotional wellbeing. Young people are invited to a single virtual group Q&A session to bring any queries after watching the videos.

The leaflets and online sessions have been developed by professionals from the Evelina, Great Ormond Street Hospital, Imperial, University College London Hospital, and the Whittington. The bite size videos and live sessions are delivered by a clinical psychologist, a dietitian, specialist nurse, occupational therapist, and physiotherapist. More complex or severely affected patients will receive one to one treatment with members of the MDT as required.

Intervention

Based on clinical expertise and theory, it is anticipated the following elements may be included in the intervention.:

* Progressive breathing pattern retraining, including education, self-observation, relaxation, body scanning, postural re-alignment
* Identifying the connections between body and mind to address anxiety and breathlessness
* Coping skills for managing anxiety using principles from narrative therapy and mindfulness
* Online materials to improve self-efficacy with home practice
* Social connection with other CYP for peer support, and resource sharing
* Activities to help CYP reconnect with their usual activities, skills, abilities, interests, support systems

DETAILED DESCRIPTION:
Hypotheses: CYP with a diagnosis of Long COVID who complete the intervention in addition to standard treatment will show a greater improvement in psychological wellbeing and demonstrate fewer functional limitations of excessive breathlessness after completing a holistic modular psychological and respiratory physiotherapy (PT) intervention compared to current standard treatment alone.

Primary objective Impact score of Strength and Difficulties (SDQ) questionnaire (included in ISARIC form - standard care assessment).

-RCADS questionnaire (17), pre- and post-intervention.

Secondary Objectives

To further answer the Ho the following measures will be taken:

* Improved dysfunctional breathing measured by multi-dimensional physiotherapy assessment of breathing pattern including Nijmegen questionnaire, breathing pattern category, SMART goal setting, lung function and cardiopulmonary exercise testing and specialist physiotherapist assessment of breathing pattern quality pre- and post-intervention.
* At baseline and 6-monthly, all CYP will complete the standard assessment questionnaires for the long COVID pan-London pathway in line with the NHSE commissioning guidance which includes the following questionnaires to assess quality of life, psychological well-being, and adaptive functioning.

  * Revised Children's Anxiety and Depression Scale (RCADS) questionnaire (17), pre- and post-intervention.
  * EQ-5D-Y (25)
  * SF-36 Quality of life (26)
  * 11-item Chalder Fatigue Questionnaire (27) and
  * Visual analogue pain scale
  * FitBit Activity monitoring including daily step counts, daily distance travelled, daily stairs climbed, sedentary minutes, low, moderate and vigorous activity minutes, sleep hours, and wear time.

Secondary research question: Are co-designed virtual psychology and physiotherapy interventions acceptable and feasible to service users?

Quantitative data: participation, attendance and dropout rates will be collected. Technical issues with being able to access the intervention will be documented.

Qualitative feedback will be obtained to enable development of the intervention.

-The facilitators will gather live feedback towards the end of each group session using a range of approaches. As part of the focus groups the CYP will review the outcome measure to get feedback if these are the things that matter to them the most. Activities to explore outcomes that matter to CYP will be reviewed in the focus groups.

Qualitative feedback will also be obtained after completion of all the group sessions when the investigator administers the post-intervention measures. This will include measures of usefulness, willingness to recommend to a friend, and qualitative questions on experience of the group, best parts of the group, and suggestions for improvement.

The investigator will also assess the impact of prior mental health problems, severity of COVID infection (community acquired vs. hospitalised) and prior functioning on intervention response.

Study Design The project is a Pan-London research project recruiting patients from across London.

The objectives of this two-part research project are firstly to co-design a novel holistic group intervention with children and young people with long COVID. The intervention will be developed based on existing literature and interventions for psychological distress and for dysfunctional breathing in similar clinical cohorts, and from focus groups with CYP with long COVID and their parents/ caregivers to ensure acceptability and appropriateness.

The second phase of this project will be to prospectively pilot the new services to assess the efficacy, acceptability, and feasibility from both the service user and service providers. The intervention will be piloted in a cohort of CYP with long COVID as an adjunctive intervention to treatment as usual, assessing impact on well being and breathing outcomes.

Phase I. Co-design Method Design and setting The intervention will be co-designed with CYP following a process informed by practice-base evidence, which centres the voices and wisdom of CYP, focuses on creativity and playfulness, and systemic and narrative approaches. The process will involve: 1) Refining the intentions of key stakeholders (including ways of bringing psychological and physiological principles into the intervention); 2) Participation of CYP; 3) Creativity and playfulness and 4) Responding to feedback (see Salvo et al., 2022).

Participation of CYP will include:

* The use of group interventions co-designed with CYP with other conditions such as diabetes, chronic pain, myalgic encephalomyelitis/chronic fatigue syndrome and medically unexplained conditions as examples to help CYP with long COVID consider some possibilities and enable them to develop their own ideas for the intervention.
* Responding to feedback and recruitment of CYP 'advisors' (name and responsibilities included in the role to be agreed with CYP)
* The use of focus groups guided by 4Pi framework and principles (NSUN, 2015) including openness and transparency about the process, finding ways to ensure the meaningful involvement of all CYP with long COVID, including those from black and minority ethnic communities, LGBTQ+ young people and other 'marginalised' groups to co-design and develop the intervention, consider recruitment and outcome measures.

The University College London Hospitals (UCLH) psychology team have developed a number of innovative and award-winning groups (20-24) that will be used as exemplars to help young people think what they might want to be included in the groups as well as delivery style (e.g., vlogs and podcasts versus leaflet), preferred frequency and length. Parents will also be invited to attend a focus group and invited to comment on similar questions. The investigators are planning to offer the groups for the CYP unaccompanied by parents.

- As part of the focus groups the CYP will review the outcome measures to get feedback if these are the things that matter to them the most. Activities to explore outcomes that matter to CYP will be reviewed in the focus groups.

Each focus group session will be via zoom and be recorded. The recording will be downloaded to a secure encrypted hospital drive. The audio recording will be used to transcribe into a script. Once this script is checked the video and audio recordings can be deleted.

Co-design participants Service Users: The investigators aim to recruit 5 to 15 young people Inclusion: CYP aged between 12-18 years old who have been referred into the Pan-London Long COVID Multi-disciplinary Team (MDT) Clinic from its inception in 2020.

Exclusion: No objective evidence of SARS-CoV-2 infection e.g., positive PCR testing or antibodies. Significant neurodevelopmental difficulties (severe autism spectrum disorder (ASD), attention deficit hyperactivity disorder (ADHD), global intellectual disability) and/or high psychiatric risk e.g., suicidality, severe emotional or behavioural dysregulation precluding participation in group intervention (PI screened during the MDT discussion and by lead researcher during telephone call for recruitment).

Phase II. Pilot Population: 40 patients (12-18 years) will be recruited from a potential pool of 214 patients referred to the pan-London long COVID MDT.

Inclusion criteria: All patients aged 12-18 years referred to the pan-London long COVID MDT with English of a standard adequate to participate in a group intervention.

Exclusion criteria: No objective evidence of SARS-CoV-2 infection e.g., positive PCR testing or antibodies. Significant neurodevelopmental difficulties (severe autism spectrum disorder (ASD), attention deficit hyperactivity disorder (ADHD), global intellectual disability) and/or high psychiatric risk e.g., suicidality, severe emotional or behavioral dysregulation precluding participation in group intervention (PI screened during the MDT discussion and by lead researcher during telephone call for recruitment).

Process: Informed consent or assent will be obtained from all CYP, and parental consent obtained for CYP under 16 years. Parents will be given access to all resources, although the intervention will be targeted towards the CYP.

Each CYP will complete a screening assessment for suitability for the trial. Once a potential participant has consented to take part they will have a Cardio-Pulmonary Exercise Test (CPET) test, lung function, 1:1 breathing pattern assessment by a respiratory physiotherapist and set up with a FitBit monitor before randomisation.

Each Fitbit will be set up by the lead researcher to a new outlook account linked to the participant number. The research team will be able to download data on daily step counts, daily distance travelled, daily stairs climbed, sedentary minutes, low, moderate and vigorous activity minutes, sleep hours, and wear time. The Fitbit will be synced to the patient's mobile phone in clinic so they can review their daily data as well. The Fitbit account will be set up with a generic date of birth, weight, and height so not to identify the patient.

CYP will be randomised (using a block randomisation approach) to receive either standard treatment or standard treatment plus intervention.

Standard treatment consists of virtual MDT discussion with referrer and advice signposting into local services for specific issues. They are sent leaflets and info on online videos (webinars) and directed to standardised information on the Your COVID Recovery Website If a patient is severely affected enough to be seen face to face, they are offered an interdisciplinary consultation, and tailored input from PT, occupational therapy (OT) and psychological services.

Access to bite size videos and leaflets and other standardised information covering the following topics: sleep, pacing, activity management, school reintegration, managing friendships, eating well and emotional wellbeing. Young people are invited to a single virtual group Q&A session to bring any queries after watching the videos/ webinars.

The leaflets have and online sessions have been developed by professionals from the Evelina, Great Ormond Street Hospital, Imperial, University College London Hospital, and the Whittington. Additional information is being developed in online video/ webinar form as the services evolve. The bite size videos/ webinars and live sessions are delivered by a clinical psychologist, a dietician, specialist nurse, occupational therapist and physiotherapist. More complex or severely affected patients will receive one to one treatment with members of the MDT as required.

Intervention

Based on clinical expertise and theory, it is anticipated the following elements may be included in the intervention:

* Progressive breathing pattern retraining, including education, self-observation, relaxation, body scanning, postural re-alignment
* Identifying the connections between body and mind to address anxiety and breathlessness
* Coping skills for managing anxiety using principles from narrative therapy and mindfulness
* Online materials to improve self-efficacy with home practice
* Social connection with other CYP for peer support, and resource sharing
* Activities to help CYP reconnect with their usual activities, skills, abilities, interests, support systems.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 12-18 years referred to the pan-London long COVID MDT with English of a standard adequate to participate in a group intervention.

Exclusion Criteria:

* No objective evidence of SARS-CoV-2 infection e.g., positive PCR testing or antibodies. Significant neurodevelopmental difficulties (severe autism spectrum disorder (ASD), attention deficit hyperactivity disorder (ADHD), global intellectual disability) and/or high psychiatric risk e.g., suicidality, severe emotional or behavioural dysregulation precluding participation in group intervention (PI screened during the MDT discussion and by lead researcher during telephone call for recruitment).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Impact score of Strength and Difficulties (SDQ) questionnaire | Through study completion, an average of 24 weeks
  25 item questionnaire comprising of 5 scales of 5 items

SECONDARY OUTCOMES:
Revised Childhood Anxiety and Depression Scale (RCADS) questionnaire | Through study completion, an average of 24 weeks
  The revised Child Anxiety and Depression Scale is a 47 item youth self reported questionnaire with subscales
EQ-5D-Y | Through study completion, an average of 24 weeks
  The EQ-5D-Y descriptive system comprises of the five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried/ sad/ unhappy
SF-36 Quality of Life | Through study completion, an average of 24 weeks
  36 item health survey - self reported quality of life measure
11 item Chandler Fatigue Questionnaire | Through study completion, an average of 24 weeks
  11 item questionnaire is divided into two components, one that measures physical fatigue and on that measures mental fatigue
Visual Analogue Scale (VAS) Pain scale | Through study completion, an average of 24 weeks
  0-10 visual analogue scale of self reported pain
FitBit Activity monitoring | Through study completion, an average of 24 weeks
  Daily step count, daily distance travelled, daily stairs climbed, sedentary minutes, low, moderate and vigorous activity minutes, sleep hours and wear time
Physiotherapy assessment of dysfunctional breathing | Through study completion, an average of 24 weeks
  Multi-dimensional physiotherapy assessment of breathing pattern
Qualitative feedback | Through study completion, an average of 24 weeks
  concurrent and retrospective feedback on the standard and new intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Brompton Hospital part of Guys and St Thomas' NHS Foundation Trust, London, Chelsea, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be handled in accordance with the Data Protection Act (2018), National Health Service (NHS) Caldecott Principles, The United Kingdom Policy Framework for Health and Social Care Research, and the condition of the Research Ethics Committee (REC) approval.
  The Case Report Forms (CRFs) will not bear the subject's name or other personal identifiable data. The subject's study Identification Number (ID) will be used for identification.
  No data will be shared with any external organisation without appropriate consent and data sharing agreement in place, as applicable.